CLINICAL TRIAL: NCT00475579
Title: Influence of an Endotracheal Tube With Polyurethane Cuff and Subglottic Secretion Drainage on Ventilator-Associated Pneumonia
Brief Title: Endotracheal Tube With Polyurethane Cuff and Subglottic Secretion Drainage
Acronym: A/N
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario de Canarias (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 01/03/2006
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Last update posted 2007-05-21 (Estimated); Status verified 2007-05

CONDITIONS: Mechanical Ventilation
Keywords: ventilator-associated pneumonia; endotracheal tube; polyurethane cuff; polyvinyl cuff; subglottic secretion drainage
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: tube with subglottic drainage and polyurethane cuff

SUMMARY:
Patients mechanically ventilated using an endotracheal tube with a subglottic secretion drainage lumen and a polyurethane cuff may develop lower ventilator-associated pneumonia than using a conventional endotracheal tube

DETAILED DESCRIPTION:
Subglottic secretions accumulated above the endotracheal cuff may progress, descending along the channels within folds of the cuff wall, to the lower respiratory tract causing VAP. Subglottic secretion drainage (SSD) appears to be effective in preventing VAP, primarily by reducing early-onset pneumonia; but it may not prevent late-onset pneumonia. We set out the hypothesis that using an endotracheal tube incorporating, besides of a subglottic secretion drainage lumen, a polyurethane cuff (which reduces channel formation and fluids leakage from the subglottic area) it should be also possible to reduce the incidence of late-onset VAP.

ELIGIBILITY:
Inclusion Criteria:

* Patients expected to require mechanical ventilation for more than 24 hours

Exclusion Criteria:

* Age <18 years,
* Pregnancy,
* HIV,
* Blood leukocytes counts <1000 cells/mm3,
* Solid or haematological tumour,
* Immunosuppressive therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2006-03; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Ventilator-associated pneumonia | 8 months

SECONDARY OUTCOMES:
Late-onset ventilator-associated pneumonia | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Lorente, MD, PhD, Principal Investigator — Intensive care unit

REFERENCES:
- [Derived] Lorente L, Lecuona M, Jimenez A, Mora ML, Sierra A. Influence of an endotracheal tube with polyurethane cuff and subglottic secretion drainage on pneumonia. Am J Respir Crit Care Med. 2007 Dec 1;176(11):1079-83. doi: 10.1164/rccm.200705-761OC. Epub 2007 Sep 13. PMID 17872488